CLINICAL TRIAL: NCT05019443
Title: WEDGES: a Prospective, Multi-center Randomized Trial for the Evaluation of Coronary Lesion Preparation With Enhanced Dilatation for Good Expansion of Stent: Assessment of a New Scoring Balloon by Quantitative Stent Enhanced Visualization
Brief Title: WEDGES: Coronary Lesion Preparation With Enhanced Dilatation for Good Expansion of Stent: Assessment of a New Scoring Balloon by Quantitative Stent Enhanced Visualization
Acronym: WEDGES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stephane Carlier (Other)
Collaborators: BrosMed Medical Co., Ltd (Industry); University of Mons (Other)
Responsible Party: Sponsor-Investigator, Stephane Carlier, Professor, University of Mons
Organization: University of Mons (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2021-08-13; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional balloon predilation (Active Comparator): the target lesion can be prepared according to standard clinical practice using SC balloons sized 0.8-1:1. Stenting using a drug-eluting stent (DES) is performed and the inflation pressure for delivery is noted, as well as the expected balloon diameter at that pressure. 2 enhanced stent imaging acquisitions (StentBoost or equivalent depending on the X-ray system used), are acquired in 2 orthogonal views. Post dilatation can be performed at operator discretion followed by a final acquisition of 2 similar orthogonal views with enhanced stent imaging. Intravascular imaging is left to the operator's discretion and is encouraged
  Interventions: Device: Conventional Balloon
- Scoring balloon predilation (Experimental): the target lesion must be prepared with a scoring balloon (SC) inflated 3 times at nominal pressure. To allow the scoring balloon to cross the lesion, it might be necessary to predilate with a small compliant balloon. The size of the scoring balloon to be used for is based on the size of the vessel. Stenting using a DES is performed and the inflation pressure for delivery is noted, as well as the expected balloon diameter at that pressure. 2 enhanced stent imaging acquisitions (StentBoost or equivalent depending on the X-ray system used), are acquired in 2 orthogonal views. Post dilatation can be performed at operator discretion followed by a final acquisition of 2 similar orthogonal views with enhanced stent imaging. Intravascular imaging is left to the operator's discretion and is encouraged
  Interventions: Device: Wedge Scoring Balloon

INTERVENTIONS:
Device: Wedge Scoring Balloon — Scoring balloon
  Arms: Scoring balloon predilation
Device: Conventional Balloon — Conventional balloon
  Arms: Conventional balloon predilation

SUMMARY:
Stent under-expansion during percutaneous coronary intervention (PCI) is one of the suboptimal results associated with a higher risk of restenosis and thrombosis. In order to obtain an optimal stent expansion, especially in lesions with calcific or fibrotic plaque, the appropriate lesion preparation before stent implantation is a crucial phase.

For this, different devices are used in everyday practices, including non-compliant balloon (NC), scoring / cutting balloons or rotational atherectomy; however, their effectiveness depends on the experience and skill of the operator. The purpose of this study is to assess the feasibility, efficacy and safety of a novel scoring balloon intended to treat calcific or fibrotic plaque of a coronary lesion

ELIGIBILITY:
Inclusion Criteria:

* Patient written consent is given A de novo lesion
* Mild to moderate burden of calcifications detected on two orthogonal views using normal radiation power

Exclusion Criteria:

* Exclusion criteria patient-related:

  1. Patient <18 years old
  2. Pregnant female
  3. Contraindication to dual antiplatelet therapy
  4. Thrombocytopenia <100 000
  5. Major surgical intervention planned

Exclusion criteria lesion-related:

1. Significant left main lesion
2. Bifurcating lesion with a significant side branch to be treated
3. Lesion length > 25 mm
4. Chronic total occlusion
5. Lesion with heavy calcifications where a rotational atherectomy or lithotripsy should be planned
6. Lesion in a graft
7. In-stent restenosis lesion
8. Lesion responsible of a STEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Stent expansion in calcified lesions assessed by stent diameter calculation using quantitative and intravascular analysis after lesion preparation using a scoring balloon is superior to conventional lesion preparation | Intravascular ultrasound (IVUS) or quantitative analysis is directly done after procedure
  The measure of stent expansion in calcified coronary lesions as assessed by quantitative coronary angiography, enhanced stent imaging and intravascular ultrasound after lesion preparation using the novel scoring semi-compliant and noncompliant balloons are superior (p<0.05) to semi compliant and non-compliant balloons.

SECONDARY OUTCOMES:
Rate of successful predilatation of calcified lesions of a scoring semi-compliant/non-compliant balloon and semi-compliant (SC)/ non-compliant (NC) balloon | Directly after procedure
Rate of residual under-expansion of stent after post-dilatation with a non-compliant balloon | Directly after procedure
Rate of procedural complication (composite of cardiac death, myocardial infarction, coronary artery perforation and cardiac tamponade) of a scoring balloon and a SC/NC balloon followed by stenting. | 1 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Carlier, Study Director — University of Mons
Locations (5):
- Belgium (5):
  - UZ Genk, Genk
  - UZ Ghent, Ghent
  - CHU Jolimont, La Louvière
  - CHU Liège, Liège
  - CHU Ambroise Paré, Mons

IPD SHARING:
Plan to Share IPD: No